CLINICAL TRIAL: NCT07203586
Title: Minimal Invasive Scoliosis or Open Surgery
Acronym: MISCOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: University of Oslo (Other); Karolinska University Hopsital (Unknown); University Hospital, Umeå (Other); Örebro University, Sweden (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other); Department of Orthopedics, Uppsala University Hospital (Unknown); Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MISCOS; 2025-01956-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2025-09-04; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Adolescent Scoliosis; Idiopathic Juvenile Scoliosis
Keywords: Idiopathic scoliosis; Minimally invasive scoliosis surgery; Traditional Open scoliosis surgical correction; Robotic assisted surgery (RAS); Win-odds; non-inferiority randomised controlled trial

STUDY DESIGN:
Intervention Model Description: Patients with idiopathic scoliosis between 10-25 years old scheduled for spinal deformity surgery will be informed about the study at the time of an outpatient visit. Patient eligibility will be established before treatment randomization. Patients will be randomized about one week prior to operation and strictly sequentially to either minimally invasive or open scoliosis surgical correction, as patients are eligible for randomization. If a patient discontinues from the study, the patient number will not be reused, and the patient will not be allowed to re-enter the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study design does not allow blinding of the surgeons and other personnel in the operating theatre. However, the patient and other health-care personnel will be blinded and held up to six months postoperatively. Patient reported outcomes will be assessed without influence of the caregiver.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive scoliosis surgery group (Experimental): Patients that will be operated by minimally invasive scoliosis surgery
  Interventions: Procedure: Minimally invasive scoliosis surgery
- Open scoliosis surgery group (Active Comparator): Patients that will be operated by traditional scoliosis surgery
  Interventions: Procedure: Traditional open scoliosis surgery group

INTERVENTIONS:
Procedure: Minimally invasive scoliosis surgery — Patients undergoing minimally invasive surgery have screws placed using the surgeon's preferred method: 3D navigation, robotic assistance, freehand, or combinations. A long incision of the skin is made without detaching the erector spinae muscles. Each screw is inserted through the musculature, and positioning is verified with intraoperative CT; misplaced screws are corrected. Rods are then shaped, placed, and deformity correction is performed. The surgeon may decorticate some or all facet joints using minimally invasive techniques before closing the wound.
  Arms: Minimally invasive scoliosis surgery group
Procedure: Traditional open scoliosis surgery group — In traditional open scoliosis surgery, the surgeon uses the preferred method for screw placement (3D navigation, robotic assistance, freehand, or combinations). A long incision is made, and the spinal musculature is detached to fully expose the posterior elements. All screws are inserted through this open area, and their positions are verified with intraoperative CT; misplacements are corrected if needed. Rods are shaped, placed, and deformity correction is performed. Decortication of facet joints, spinous processes, and laminae may be performed with a high-speed burr or similar technique. The wound is then closed.
  Arms: Open scoliosis surgery group

SUMMARY:
Surgical treatment for idiopathic scoliosis usually involves open surgery from the back (posterior approach). This method corrects the curve and stabilizes the spine using screws and rods, followed by a fusion of the treated segments. The goal is to achieve the best possible alignment of the spine.

This type of surgery can be demanding for the body and often requires a longer hospital stay because of tissue damage and pain after the procedure. Traditionally, patients stayed in the hospital for up to a week or more.

In recent years, recovery programs such as ERAS (Enhanced Recovery After Surgery) have been introduced. These programs include better pain control, faster mobilization, and improved preparation before surgery. Thanks to these improvements, many patients can now go home one to two days after surgery instead of several days.

There has also been a development of minimally invasive surgery (MIS) techniques in spine surgery. These techniques aim to reduce tissue damage and blood loss compared to traditional open surgery. Smaller incisions can lead to less scarring, less pain, and potentially faster recovery. Because scoliosis surgery is complex, it is important to study whether MIS offers the same safety and benefits as traditional surgery.

Minimally invasive surgery makes correct screw placement in the curved spine more challenging, as the usual anatomical landmarks are not fully exposed. To ensure accuracy, MIS often uses advanced technologies such as intraoperative 3D imaging or robotic-assisted surgery (RAS).

The purpose of this project is to evaluate whether MIS is as safe and effective as traditional open surgery. The study will compare both methods regarding the need for additional surgery, complications, infections, pain, and bone fusion after surgery. It will also examine hospital stay, degree of curve correction, accuracy of screw placement, changes in nerve function during surgery, blood loss, operation time, and patient-reported outcomes.

Most existing studies on MIS in scoliosis are based on older or small patient series, and randomized controlled trials are lacking. This research will provide scientific evidence to guide future treatment choices. The aim is to determine whether MIS can deliver the same correction and safety as open surgery while reducing pain, blood loss, and recovery time. If proven effective, these techniques could improve recovery and quality of life for many scoliosis patients.

DETAILED DESCRIPTION:
1. Purpose and Aims:

   The primary aim of this study is to evaluate the effectiveness of minimally invasive surgery (MIS) compared to traditional open surgery for the treatment of idiopathic scoliosis. While open surgery remains the gold standard for spinal correction, it is associated with significant tissue trauma, extended hospitalization, and postoperative pain. The emergence of MIS techniques offers potential benefits, including reduced tissue damage, shorter hospital stays, and faster recovery. However, the long-term outcomes and efficacy of MIS in scoliosis correction remain unclear due to the lack of high-quality evidence, particularly from randomized controlled trials (RCTs).

   This study is designed as a multi-center, two-arm, non-inferiority RCT to determine whether MIS can achieve comparable outcomes to open surgery in terms of:
   1. Primary surgical outcomes: Reoperation rates, serious complications, surgical site infections, postoperative pain levels, and fusion success.
   2. Secondary measures: Hospitalization duration, screw placement accuracy, neurophysiological events, blood loss, operative time, and patient-reported outcomes (PROMs).

   A key challenge in MIS is the accurate placement of implants in the deformed spine while minimizing disruption to surrounding tissues. The study will assess whether the use of intraoperative 3D imaging and robotic-assisted surgery (RAS) enhances precision while maintaining surgical success.

   By addressing these critical questions, this trial aims to provide high-quality evidence on the role of MIS in scoliosis treatment. If MIS proves to be as effective as open surgery while offering faster recovery and fewer complications, it could lead to a paradigm shift in scoliosis management, improving patient care and reducing healthcare burden.
2. Background:

   Idiopathic scoliosis is the most common spinal deformity, affecting 1.9-3.0% of the population and often requiring extensive surgical treatment during youth. Beyond the challenges of treatment and the high healthcare costs, scoliosis can significantly impact quality of life, both in adolescence and adulthood. Surgical intervention is typically indicated for Cobb angles exceeding 45 degrees in skeletally immature- and 50 degrees in skeletally mature patients. The standard approach involves posterior spinal fusion via open surgery, allowing near-anatomical correction but resulting in extensive tissue damage, prolonged hospitalization, and significant postoperative pain. Recent protocols such as Enhanced Recovery After Surgery (ERAS) have optimized pain management, enabling some patients to be discharged within 1-2 days.

   Minimally invasive surgery (MIS) has evolved in spine surgery, offering potential advantages such as reduced tissue trauma, lower blood loss, and faster recovery. However, its role in scoliosis surgery remains uncertain, particularly regarding its ability to achieve the same level of deformity correction and spinal fusion success as open surgery. One key challenge in MIS is accurate implant placement in a deformed spine while minimizing tissue disruption and preserving anatomical landmarks. This has led to the integration of intraoperative 3D imaging and robotic-assisted surgery (RAS) to enhance screw placement accuracy.

   To date, most evidence on MIS in scoliosis surgery comes from retrospective and observational studies, with a lack of randomized controlled trials (RCTs). While MIS has rapidly developed in the field of degenerative spine surgery, it is important to investigate whether MIS in patients with idiopathic scoliosis is non-inferior than traditional open surgery and at the same time not compromise other factors of a "successful" operation such as the degree of correction and fusion.
3. Study design:

   a. Research questions The primary objective of this project is to assess whether minimally invasive surgery (MIS) is non-inferior to traditional open surgery in terms of reoperation rates, serious complications, surgical site infections, pain, and fusion success in the long term. Additionally, the investigators aim to compare the two techniques regarding hospitalization time, screw placement accuracy, neurophysiological events, blood loss, operative time, and patient-reported outcome measures (PROMs).

   A randomized controlled trial (RCT) will be conducted to minimize selection bias and systematically evaluate the advantages and limitations of MIS compared to open surgery in scoliosis correction. The study follows a pragmatic approach, utilizing existing surgical techniques and infrastructures, including established MIS techniques, navigation systems, hospital and quality registries, and imaging systems. Randomization will be performed within the Swespine registry platform or RedCap.

   Definition of MIS: The technique preserves the posterior spinal musculature by avoiding detachment from the spinous processes and laminae, except where necessary for screw insertion. Surgeons may use either a single long incision or multiple short incisions, ensuring muscle-sparing principles while achieving spinal stabilization.

   b. Variables and measures

   The primary endpoint is the assessment of a group of variables by the statistical method of "win odds". The variables are in hierarchic order:

   i. No reoperations at 2 years after surgery. A reoperation is defined as a secondary surgical procedure related to the index procedure and involving the spine after the index procedure.

   ii. No serious complication related to the procedure. Serious complication is defined as a life-threatening complication or a complication related to substantial invalidity.

   iii. No early surgical site infection (SSI) that is defined with onset up to 12 weeks postoperatively.

   iv. No other infection related to the inpatient stay like pneumonia or urinary tract infection (UTI).

   v. Assessment of pain at 2 years follow-up: The numeric rating scale (NRS) for back and leg pain, respectively will be used measured on a scale from 0 (no pain) to 10 (worst possible pain). Data will be collected from Swespine or similar platforms.

   vi. The SRS-22r is a scoliosis specific questionnaire aiming to estimate quality of life in patients with scoliosis. It covers function, pain, self-image, mental health, and satisfaction.

   vii. Radiologically healed fusion at 2 years f-u. A radiologically healed fusion is defined as bone bridging along the originally operated levels. A vertebral segment will be considered fused if one or both of the following conditions is satisfied:

   a. Bone bridge over at least one facet joint b. Bone bridge between the vertebral bodies The following secondary objectives will be studied in comparisons between MIS and open operating procedures.

   i. Inpatient stay in days. ii. Total procedure time normalized to number of spinal levels. iii. Perioperative blood loss (in mL). iv. Postoperative pain relief assessed by NRS at discharge. Additionally, given and prescribed doses of analgesics will be registered from the hospital files.

   v. Health economics: Total cost per patient during the first 2 years of the study including cost of possible re-admissions and reoperations related to index surgery.

   vi. Accuracy at first attempt: Screws that are not placed and screws that are placed but repositioned after intraoperative verification are noted in the protocol.

   vii. Technical accuracy of screw placement at 2 years follow-up. An accurately placed screw is defined as of grade Ia and Ib according to Heintel classification.

   viii. Intraoperative neurophysiological monitoring. Motor evoked potential, sensory evoked potential and electromyography data will be collected to investigate any changes in neurophysiological parameters. Any deviations will be noted.

   ix. Patient reported outcome measures (PROMS) c. Patient selection Patients between 10-25 years old scheduled for spinal deformity surgery will be informed about the study at the time of an outpatient visit. Patient eligibility will be established before treatment randomization. Patients will be randomised preoperatively and strictly sequentially, as patients are eligible for randomisation. If a patient discontinues from the study, the patient number will not be reused, and the patient will not be allowed to re-enter the study.

   Inclusion criteria:

   (i) Written informed consent, (ii) idiopathic scoliosis, (iii) age between 10-25 years, (iv) posterior correction for scoliosis, (v) normal walking ability, (vi) major curve Cobb angle 75 or less.

   Exclusion criteria:

   (i) inability to give informed consent, (ii) other diagnosis of scoliosis than "idiopathic", (iii) rigid curves that require posterior or three-column osteotomy/ies, (iv) previous surgery at the operated levels, (v)BMI > 35, (vi) psychological factors that make the patient unsuitable for inclusion in the study (e.g., substance abuse, developmental disability).

   d. Estimated sample size and power In order to use the win-odds method for a non-inferiority study the investigators performed more than 1000 simulations using the statistical software R. The primary variables listed in 6.1 were used to calculate the sample size and assumed that the outcomes are independent and that the outcomes were equally distributed among study arms (i.e. the investigators simulated a win-odds of 1.0). The power of the study was set to 80% with a lower limit of confidence interval for win-odds (also called non-inferiority limit) to above 0.60 and calculated a sample size of 150 individuals divided into two treatment arms. The possible number of dropouts until the 2-year follow-up was set to 20%, and the total sample size therefore adjusted to 180 individuals.

   The non-inferiority limit is the probability of a patient in the active arm (minimally invasive procedure) to win over a control patient given an evenly distributed number of ties.

   In the case that the MIS group shows slight benefits compared to the open surgery group then the non-inferiority limit will shift towards 1.0 as the win odds will be greater than 1.0 which was assumed in the sample size simulation.

   e. Statistical methods

   Primary variables:

   The investigators selected the above described seven variables in hierarchic order to conduct a win-odds analysis. The variables were selected based on the clinical impact that they have on the patient. The method of win-odds was first introduced as win-ratio in order to analyze composite endpoints based on clinical priorities. The method compares each treatment subject to all controls and the outcome is registered as "win", "lose" or "tie". In order to handle large numbers of ties the win-odds was introduced that assigns 50% of the ties to both the numerator and the denominator. Particularly in non-inferiority trials the use of win-odds instead of win-ratio may be more suitable since ties in non-inferiority studies may represent a comparable treatment effect and their number is substantial.

   Secondary variables For the secondary variables descriptive statistics will be used to characterize the data; means and 95% confidence intervals will be used for parametric data, medians and interquartile ranges for non-parametric data, and number (proportions) for categorical data. Data from the different groups will be compared based on the 'intention to treat' principle. Statistical expertise blinded for treatment allocation will perform the statistical analyses.

   f. Feasibility The Akademiska hospital in Uppsala performs approximately 80 spine deformity surgeries yearly and it is estimated that 1/4 of these meet the inclusion criteria for the study. Similar estimations are done for the rest of the centers with a total enrolment of approximately 50 patients per year. Our time plan includes study start (mid 2025), last patient included (2028) and last 2 year follow up (2029). Registry outcome data are collected preoperatively, at 1 year and 2 years. Registry data may also be collected at 5 and 10 years.

   A total of eight pilot cases has been already performed in Akademiska hospital during 2024 and early 2025 with satisfactory correction rate and a normal expected postoperative follow-up.

   g. Risk mitigation Since surgical intervention is the established standard of care, the investigators consider it ethically justifiable for research participants to be exposed to the inherent risks of the procedure.

   Minimally invasive surgical (MIS) techniques are already widely used in degenerative spine surgery and spinal trauma, where they are well-established and have demonstrated favorable outcomes. With this study, the investigators aim to evaluate and apply MIS for the treatment of idiopathic scoliosis.

   Two potential risks theoretically associated with MIS in scoliosis surgery are:

   i. Achieving optimal anatomical correction of scoliosis may be more challenging compared to traditional open surgery.

   ii. Bone fusion in the MIS group may be inferior to that in the open surgery group.

   iii. If a technical problem with the 3D/navigation system or RAS system is encountered during surgery, the patient will be kept in the group to which he or she was randomized. This means that a possible MIS approach needs to be converted to open technique to enable screw placement by free hand technique. The patient will remain in the group to which he or she was randomized to and will not be replaced.

   Despite these potential risks, the investigators believe it is essential to scientifically investigate the use of MIS in scoliosis patients. MIS has the potential to offer significant advantages, including fewer reoperations, faster rehabilitation, lower infection rates, reduced blood loss, and shorter hospital stays. The knowledge gained from this study could contribute to improved treatment strategies and enhanced quality of life for patients with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Idiopathic scoliosis
* Age between 10-25 years
* Planed surgery: Posterior correction for scoliosis
* Major curve Cobb angle 75 degrees or less

Exclusion Criteria:

* Inability to give informed consent
* Other diagnosis of scoliosis than "idiopathic"
* Rigid curves that require posterior or three-column osteotomy/ies
* Previous surgery at the operated levels
* BMI > 35
* Psychological factors that make the patient unsuitable for inclusion in the study (e.g., substance abuse, developmental disability)

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the assessment of a composite group of variables by the statistical method of "win odds". The variables are listed in hierarchic order in the "description" below. | From the inclusion of the first subject up to two years after the operation of the last subject.
  The composite primary endpoint includes: (i) no reoperation within two years (defined as any secondary spinal procedure related to the index operation); (ii) no serious complications, defined as life-threatening events or complications associated with long-term disability; (iii) absence of early surgical site infection, defined as infections occurring within 12 weeks postoperatively; (iv) absence of other inpatient-related infections, such as pneumonia or urinary tract infections; (v) patient-reported pain at two years, measured using the Numeric Rating Scale (NRS) for back and leg pain; (vi) quality of life assessed with the SRS-22r questionnaire, which captures dimensions such as pain, function, self-image, mental health, and satisfaction; and (vii) radiological evidence of successful spinal fusion, defined as bone bridging across the operated spinal levels, either through the facet joints or between vertebral bodies.

SECONDARY OUTCOMES:
Inpatient stay | During the discharge of each subject, assessed up to two weeks after the operation of the last subject.
  Inpatient stay from the day of operation up to discharge measured in days
Deformity correction rate | The assessment will take place during the first follow up of each subject (three months postoperatively) and will be assessed up to the first follow-up of the last subject.
  The deformity correction rate will be assessed as Cobb-angle correction in a postoperative x-ray from the first standing radiograph compared to the last preoperative radiograph. The correction of the curve will be calculated according to the formula: (preoperative Cobb angle - postoperative Cobb angle) / (preoperative Cobb angle) × 100%.
Progression of Cobb angle in the operated levels at 2-years standing x-ray | At 2-year follow-up for each subject assessed up to the 2-year follow-up of the last subject.
  Progression of Cobb angle in the operated levels at 2-years standing x-ray compared to the 3-month (first follow-up) x-ray. The progression of the curve will be calculated according to the formula: (2-year Cobb angle - 3-month Cobb angle) / (2-year Cobb angle) × 100%.
Progression of secondary curve angles at 2-years standing x-ray | During the 2-year follow-up for each subject up to the 2-year follow-up of the last subject.
  Progression of secondary curve angles at 2-years standing x-ray compared to the 3-month (first follow-up) x-ray. The progression of the curve will be calculated according to the formula: (2-year Cobb angle - 3-month Cobb angle) / (2-year Cobb angle) × 100%.
Perioperative blood loss | Assessed during the surgery of each subject
  Perioperative blood loss in mL
Accuracy of screw placement at the first attempt | Assessed during the surgery of each subject.
  Accuracy of screw placement will be assessed as a score, calculated as the number of correctly placed screws divided by the total number of screws specified in the preoperative plan (see Appendix 1 in the study protocol). The maximum score is 1, indicating perfect placement according to the preoperative plan. Screws graded Ia or Ib by the Heintel classification (see reference list) are defined as correctly placed. Screws that are not inserted, or that require repositioning after intraoperative verification, will be recorded in the protocol and classified as NOT correctly placed.
Total procedure time | From the start until the end of surgery for each subject.
  Operation time in minutes normalised to the number of spinal levels from the upper to the lower instrumented vertebra.
Intraoperative neurophysiological monitoring | During the surgery of each subject.
  Neurophysiological monitoring is always performed as routine during spinal deformity surgery, with the exception of patients that are non-ambulatory. Motor evoked potential, sensory evoked potential and electromyography data will be collected to investigate any changes in neurophysiological parameters. Any deviations will be noted.
Health economics | From the discharge of the first subject up to two years from the discharge of the last subject
  Total cost per patient during the first 2 years of the study including cost of possible re-admissions and reoperations related to index surgery. Data on costs on the individual level will be collected. These consist of costs for the inpatient and outpatient visits (including surgery, radiographs, navigation), analgesic and antibiotic treatments as well as possible re-admissions related to index surgery.
SRS-22r | Patient reported outcome measure (PROM) registered in Swespine registry or similar platforms 1, 2, 5 and 10 years postoperatively.
  The SRS-22r is a scoliosis specific questionnaire aiming to estimate quality of life in patients with scoliosis. It contains 24 items divided into 5 domains covering function, pain, self-image, mental health, and satisfaction. An index value is calculated for each domain and a total index value is possible to calculate ranging from 1 (worst) to 5 (best).
EOSQ-24 | Patient reported outcome measure (PROM) registered in Swespine registry or similar platforms 1, 2, 5 and 10 years postoperatively.
  EOSQ-24 is a proxy answered questionnaire and will be used in individuals up to the age of 15. It consists of 24 questions of daily function, pain, pulmonary function and mobility [see reference list]
Oswestry Disability index (ODI) | Patient reported outcome measure (PROM) registered in Swespine registry or similar platforms 1, 2, 5 and 10 years postoperatively.
  Oswestry Disability index (ODI) is used in individuals from 15 years and older. ODI is a back specific index measuring disability due to back pain [see reference list]. It is the recommended instrument for studies concerning back pain. An index from 0-100 is calculated. An ODI of 0-20 indicate minimal disability, 21-40; moderate disability, 41-60; severe disability, 61-80; severely crippled, 81-100; bed-bound.
EQ-5D 3 level | Patient reported outcome measure (PROM) registered in Swespine registry or similar platforms 1, 2, 5 and 10 years postoperatively.
  EQ-5D 3 level is a generic quality of life instrument and consists of five areas reflecting mobility, self-care, usual activities, pain/discomfort and anxiety/depression [see reference list]. Response aternatives range from no problems to extreme problems. An index can be calculated and depending on baseline value set used the index runs between approximately -0.5 (worst possible health) to 1.0 (best possible health). The EQ-5D-3L will be used for health economic analyses. The EQ-VAS is part of the EQ-5D and registers the patient's self-rated health on a visual analogue scale (from 0 to 100; best).
Postoperative pain relief | The information will be given by each subject at discharge as well as registered in Swespine registry or similar platforms 1, 2, 5 and 10 years postoperatively.
  Assessed by Numeric Rating Scale (NRS) for back and leg pain, respectively, and is measured on a scale from 0 (no pain) to 10 (worst possible pain). Additionally, given and prescribed doses of analgesics that follow clinical routine protocols will be registered from the hospital files.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Schizas, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Akademiska University hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual data cannot be shared according to Swedish law. However, aggregated data, and completely deidentifed data that can be shared without the possibility to track the data to an individual may be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol, statistical analysis and informed consent form is currently available upon request from the study coordinator. The complete clinical study report will be available upon request after the 2-year follow-up of the last subject included. Data registered in Swespine or similar platforms are available upon request.
Access Criteria: The principal investigator and study coordinators will have access to the data. Other researchers can have access to supporting information upon request.

REFERENCES:
- [Background] Dong G, Huang B, Chang YW, Seifu Y, Song J, Hoaglin DC. The win ratio: Impact of censoring and follow-up time and use with nonproportional hazards. Pharm Stat. 2020 May;19(3):168-177. doi: 10.1002/pst.1977. Epub 2019 Oct 31. PMID 31671481
- [Background] Pocock SJ, Ariti CA, Collier TJ, Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. Eur Heart J. 2012 Jan;33(2):176-82. doi: 10.1093/eurheartj/ehr352. Epub 2011 Sep 6. PMID 21900289
- [Background] Peng L. The use of the win odds in the design of non-inferiority clinical trials. J Biopharm Stat. 2020 Sep 2;30(5):941-946. doi: 10.1080/10543406.2020.1757690. Epub 2020 May 31. PMID 32475213
- [Background] Burstrom K, Johannesson M, Diderichsen F. Swedish population health-related quality of life results using the EQ-5D. Qual Life Res. 2001;10(7):621-35. doi: 10.1023/a:1013171831202. PMID 11822795
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Matsumoto H, Williams B, Park HY, Yoshimachi JY, Roye BD, Roye DP Jr, Akbarnia BA, Emans J, Skaggs D, Smith JT, Vitale MG. The Final 24-Item Early Onset Scoliosis Questionnaires (EOSQ-24): Validity, Reliability and Responsiveness. J Pediatr Orthop. 2018 Mar;38(3):144-151. doi: 10.1097/BPO.0000000000000799. PMID 27299779
- [Background] Heintel TM, Dannigkeit S, Fenwick A, Jordan MC, Jansen H, Gilbert F, Meffert R. How safe is minimally invasive pedicle screw placement for treatment of thoracolumbar spine fractures? Eur Spine J. 2017 May;26(5):1515-1524. doi: 10.1007/s00586-016-4908-3. Epub 2016 Dec 8. PMID 27933475
- [Background] Danielsson AJ, Romberg K. Reliability and validity of the Swedish version of the Scoliosis Research Society-22 (SRS-22r) patient questionnaire for idiopathic scoliosis. Spine (Phila Pa 1976). 2013 Oct 1;38(21):1875-84. doi: 10.1097/BRS.0b013e3182a211c0. PMID 23846501

DOCUMENTS (1):
  • Study Protocol (2025-09-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT07203586/Prot_000.pdf